CLINICAL TRIAL: NCT00934284
Title: Effectiveness of Physical Therapy As an Adjunct to a Selective Nerve Root Block in the Treatment of Lumbar Radicular Pain from Disk Herniation
Brief Title: Effectiveness Study of Physical Therapy As an Adjunct to a Lumbar Therapeutic Selective Nerve Root Block
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Anne Thackeray, PhD, University of Utah
Other Study IDs: 00014476
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Sciatic Neuropathy; Radiculopathy; Intervertebral Disk Displacement
Keywords: sciatic neuropathy; physical therapy; spinal injections
MeSH Terms: conditions — Sciatic Neuropathy; Radiculopathy; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Injection only: Participants receive a therapeutic selective nerve root block and advice to return to normal activity as tolerated.
  Interventions: Other: Lumbar injection
- Injection plus physical therapy: Participants are referred to physical therapy within one week of receiving a therapeutic selective nerve root block. Physical therapy consists of end-range movements in a directional preference and/or mechanical traction to reduce radicular symptoms.
  Interventions: Other: Rehabilitation following lumbar injection

INTERVENTIONS:
Other: Lumbar injection — Patients are instructed to resume normal activity as tolerated.
  Groups: Injection only
Other: Rehabilitation following lumbar injection — Participants are referred to an average of four weeks of physical therapy after receiving a lumbar injection. Physical therapy designed to include end-range directional preference exercises and/or mechanical traction to reduce lower extremity symptoms and progress activity tolerance.
  Groups: Injection plus physical therapy

SUMMARY:
The purpose of this study is to determine if participation in physical therapy in conjunction with a selective nerve root block in the lumbar spine is more effective than just receiving the injection alone for patients with low back and leg pain from a disk herniation (sciatica).

DETAILED DESCRIPTION:
Recent reviews report moderate to strong evidence for short-term relief but limited evidence for long-term improvement. Anecdotal reports and case studies suggest good outcomes with various physical therapy interventions however well-designed research studies examining treatments in combination are lacking. The management of lumbar radicular pain often includes the combination of physical therapy and therapeutic selective nerve root blocks with the rationale that reducing inflammation and pain will permit greater participation in physical therapy. The effectiveness of this combination of treatment has not been studied and is the purpose of this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* MRI evidence of disk herniation in the lumbar spine consistent with clinical presentation
* Pain and/or paresthesia in the lumbar spine and a distribution extending distal to the gluteal fold within 24 hours of enrollment
* Scheduled to receive a therapeutic selective nerve root block

Exclusion Criteria:

* Any lumbar surgery within six months of the baseline examination
* Any prior lumbar surgery involving fusion
* Medical red flags indicating a serious pathology such as neoplasm, infection, or fracture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with low back pain, with clinical and imaging findings consistent with lumbar disk herniation, and scheduled to receive a selective nerve root block.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry Disability Index | Baseline (pre-injection), 8 weeks (post-injection), 6 months post-injection

SECONDARY OUTCOMES:
Global Rating of Change | 8 weeks (post-injection) and 6 months (post-injection)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, Principal Investigator — Associate Professor
Locations (1):
- Intermountain Healthcare, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Thackeray A, Fritz JM, Brennan GP, Zaman FM, Willick SE. A pilot study examining the effectiveness of physical therapy as an adjunct to selective nerve root block in the treatment of lumbar radicular pain from disk herniation: a randomized controlled trial. Phys Ther. 2010 Dec;90(12):1717-29. doi: 10.2522/ptj.20090260. Epub 2010 Sep 23. PMID 20864600